CLINICAL TRIAL: NCT05833152
Title: Correlation Analysis of Knee Extension Lag Angle and Knee Function After Total Knee Arthroplasty
Brief Title: Correlation Between Preoperative Knee Extension Lag and Functional Outcome After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022846
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2023-05

CONDITIONS: Extension Lag; Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- <5°
  Interventions: Procedure: total knee arthroplasty
- 5-10°
  Interventions: Procedure: total knee arthroplasty
- 10-15°
  Interventions: Procedure: total knee arthroplasty
- ≥15°
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — To observe the postoperative functional outcome of patients with knee extension lag at different angles

SUMMARY:
To explore the relationship between different knee extension hysteresis angles and functional outcome of knee joint after total knee replacement

DETAILED DESCRIPTION:
1. Collect perioperative baseline data

   Subjects were recruited and perioperative baseline data were collected: ① Demographic information, including age, sex, height, weight, affected knee, etc. ②Body structure and function: joint motion, knee extension hysteresis angle, pain NRS, WOMAC assessment, and ultrasonic knee extension mechanism were measured before and 3 days after surgery.
2. Postoperative follow-up

   The patients were followed up for 3 months, and 6 weeks /3 months after surgery was selected as the follow-up node. The follow-up included postoperative range of motion, knee extension hysteresis Angle, pain NRS, WOMAC assessment, ultrasonic measuring knee extension mechanism, TUG Test (Timed Up-to-go Test), isometric muscle force test, balance postural graph, gait analysis, etc.
3. Data analysis

   1. Multi-factor regression analysis was performed to determine the main outcome indicators of WOMAC evaluation at 3-month follow-up, including range of motion, Angle of knee extension hysteria, pain NRS, ultrasonic knee extension device, TUG Test (Timed Up-to-go Test), isoktatic muscle force test, balance postural graph and secondary outcome indicators of gait analysis. The perioperative knee extension hysteresis Angle was used as the independent variable to construct the postoperative regression model of knee function.
   2. According to the Angle of knee extension hysteresis in perioperative period, patients were divided into 4 groups: ≤5°, 5-10°11-15°, ≥15°, The results of range of motion, knee extension hysteresis Angle, pain NRS, WOMAC score, ultrasonic knee extension device, TUG Test (Timed Up to go Test), iso-tachykinesis test, balance postural mapping and gait analysis were compared among all groups 3 months after surgery.
4. Study outcome

Follow-up was completed; The patient underwent revision surgery for knee osteoarthritis. The patient dropped out of the trial for personal reasons; Other unforeseen circumstances prevented the patient from continuing the trial.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who meet the diagnostic criteria of knee osteoarthritis (age >45 years old); (2) Patients admitted to the Department of Orthopedics of the Third Hospital of Beijing Medical University and preparing to receive TKA surgery; (3) The patient has good cognitive function and good compliance, and can cooperate with various examinations; (4) Voluntarily participate in the study and sign the informed consent;

Exclusion Criteria:

* (1) Patients with lower extremity fracture and severe lumbar spinal stenosis that affect postoperative functional recovery; (2) Patients with severe cerebrovascular disease who cannot cooperate with postoperative rehabilitation exercise; (3) The time interval of double knee replacement was less than 3 months.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Orthopaedics of Peking University Third Hospital for total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
WOMAC | three months after surgery
  Knee functional scale

SECONDARY OUTCOMES:
Thickness of vastus medialis muscle | three months after surgery
  muscle thickness
range of motion | three months after surgery
  Reflect knee function

CONTACTS AND LOCATIONS:
Overall Officials: Yang yanyan, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGinn TL, Etcheson JI, Gwam CU, George NE, Mohamed NS, Mistry JB, Ananaba U, Bhave A. Short-term outcomes for total knee arthroplasty patients with active extension lag. Ann Transl Med. 2018 Jun;6(11):204. doi: 10.21037/atm.2018.05.38. PMID 30023367